CLINICAL TRIAL: NCT05403060
Title: Educational Nutritional Intervention to Increase the Consumption of Vegetables and Fruits and Decrease the Consumption of Ultra-processed Foods in Adolescents: Randomized Controlled Trial by Conglomerates
Brief Title: Educational Nutritional Intervention for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Gabriela Macedo Ojeda, PhD in Public Health Sciences, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-88
Record Dates: First submitted 2022-02-24; First posted 2022-06-03 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Early Intervention, Educational; Health Promotion; Feeding Behavior; Adolescent Health
Keywords: Vegetables; Fruit; Ultra-processed Food
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: An intervention group and a control group (no intervention, with usual education)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Educational nutritional intervention, based on the Social Cognitive Theory
  Interventions: Behavioral: ALIADA: Alimentación, Adolescencia y Ambiente
- Control (No Intervention): Regular school education, without educational nutritional intervention

INTERVENTIONS:
Behavioral: ALIADA: Alimentación, Adolescencia y Ambiente — The objective of the educational nutritional intervention is to promote in adolescents an increase in their consumption of vegetables and fruits and a decrease in their consumption of ultra-processed foods, through the application of the TSC constructs, with the use of education by pairs as the main strategy (peer leaders). It lasts two months, includes three exclusive sessions for peer leaders and five sessions for all participants, where the leaders, together with the researchers, will lead the activities of the sessions, as well as a general event for all high school students. Intervention activities include: electronic presentations, videos, food preparation and label reading workshops, individual and team reflection activities, goal setting and monitoring, board games, contests, among others. In addition, each participant is given a workbook, which contains key messages and activities for each educational session.
  Arms: Intervention

SUMMARY:
Randomized controlled trial by conglomerates whose objective is to evaluate the effectiveness of an educational nutritional intervention, based on the Social Cognitive Theory, for the increase in the consumption of vegetables and fruits and the decrease in the consumption of ultra-processed foods in adolescent high school students, in the University of Guadalajara, in Guadalajara, Jalisco.

DETAILED DESCRIPTION:
Background: Adolescent nutrition is of vital importance for their growth and development, at this stage eating habits for adult life are consolidated. However, currently the eating habits of adolescents are mainly characterized by a high consumption of ultra-processed foods and a low consumption of vegetables and fruits. Effective nutritional interventions focused on this age group can contribute to the prevention of adolescent diseases at the current stage and in later stages.

Objective: To evaluate the efficacy of an educational nutritional intervention, based on the Social Cognitive Theory, to increase the consumption of vegetables and fruits and decrease the consumption of ultra-processed foods, in adolescent high school students at the University of Guadalajara (UDG), in Guadalajara, Jalisco, in the year 2022.

Material and methods: Randomized controlled trial by conglomerates, students from the school groups chosen at random, from two high schools (one as a control group and another intervention) also chosen at random will be included. Adolescents who agree to participate will complete pre- and post-intervention assessments on fruit and vegetable consumption and ultra-processed foods. A multilevel analysis will be used to compare post-intervention variables between groups.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the included high schools (1st to 6th semester, morning and evening shift)
* That they agree to participate and complete the assent and informed consent form

Exclusion Criteria:

* Students who do not wish to participate

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Change in vegetables and fruits | 2 months
  Pre-post intervention change in vegetable and fruit consumption (servings/day (direct values, no scores assigned), post intervention consumption minus pre intervention consumption, as measured by a semiquantitative food frequency questionnaire, positive values of change are desirable , that is, increased consumption of vegetables and fruits)
Change in ultra-processed foods | 2 months
  Pre-post intervention change in consumption of ultra-processed foods (servings/day (direct values, no scores assigned)), post intervention consumption minus pre intervention consumption, as measured by a semiquantitative food frequency questionnaire, negative values of change are desirable, that is, reduction in the consumption of ultra-processed foods)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Macedo Ojeda, PhD, Study Director — Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara
Locations (1):
- Upper Secondary Education System of the University of Guadalajara, Guadalajara, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McAlister AL, Perry CL, Parcel G. How individuals, environments and health behavior interact: social cognitive theory. In: Glanz K, Rimer BK, Viswanath K, eds. Health Behavior and Health Education: Theory, Research and Practice. 4°. Jossey-Bass A Wiley Imprint; 2008:169-188.
- See also: Encuesta Nacional de Salud y Nutrición 2018 — http://ensanut.insp.mx/encuestas/ensanut2018/doctos/informes/ensanut_2018_presentacion_resultados.pdf